CLINICAL TRIAL: NCT00395538
Title: Effects of PTH Replacement on Bone in Hypoparathyroidism
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pharmacy temporarily suspended by FDA
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070016; 07-D-0016
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hypoparathyroidism; DiGeorge Syndrome
Keywords: Parathyroid; Bone Biopsy; Calcium-Sensing Receptor; Bone Density; Bone Turnover; Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism; DiGeorge Syndrome | interventions — Parathyroid Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Biopsy (Other): Subjects are randomized to have the second bone biopsy done 1,2, or 4 years after the start of PTH.
  Interventions: Drug: PTH 1-34

INTERVENTIONS:
Drug: PTH 1-34 — Given twice daily by subcutaneous
  Other Names: HPTH

SUMMARY:
Hypoparathyroidism is a rare condition associated with a low level of parathyroid hormone (PTH) in the blood. Hypoparathyroidism can be genetic and show up in childhood, or it can occur later in life. If it occurs later, it is usually due to damage or removal of the parathyroid glands during neck surgery. PTH helps control the amount of calcium in blood, kidneys, and bones. Low levels of calcium in the blood can cause a person to feel sick. It can cause cramping or tingling in the hands, feet, or other parts of the body. A very low blood calcium can cause fainting or seizures.

The standard treatment for hypoparathyroidism is a form of vitamin D (calcitriol) and calcium supplements. Keeping normal blood levels of calcium can be difficult. Sometimes there is too much calcium in the urine even if the calcium levels in the blood are low. High calcium in the kidneys and urine can cause problems such as calcium deposits in the kidney (nephrocalcinosis) or kidney stones. High levels of calcium in the kidney may keep the kidney from functioning normally. Treatment with PTH will replace the hormone you are missing. Your disease may be better controlled on PTH than on calcium and calcitriol.

Researchers at the NIH have conducted prior studies to establish synthetic human parathyroid hormone 1-34 (HPTH) as a treatment for hypoparathyroidism. Other studies have shown that PTH may improve calcium levels in blood and urine. The primary purpose of this research study is to evaluate the effects of synthetic human parathyroid hormone 1-34 (HPTH) replacement therapy on bone in adults and teenagers with hypoparathyroidism.

The study takes 5 (Omega) years to complete and requires 12 inpatient visits to the National Institutes of Health Clinical Center in Bethesda, MD. The first visit will help the study team decide whether you are eligible. This visit will last 2 to 3 days. After taking calcium and calcitriol for 1 - 7 months you will return to the NIH Clinical Center for the baseline visit. The baseline visit is the visit that you will start your PTH; you will also undergo a bone biopsy during the visit. The baseline visit may last 7 to 10 days. You will then take PTH twice a day for 5 years. You will be asked to return to the NIH clinical center every 6 months for 10 follow-up visits. During one of the follow-up visits, you will have a second bone biopsy taken from the other hip. That second biopsy will be done after 1 year, 2 years, or 4 years of taking PTH; the researchers will assign the timing of the second biopsy randomly. You will be asked to go to your local laboratory for blood and urine tests between each follow up visit. At first the blood tests will occur at least once a week. Later, you will need to go to your local laboratory for blood tests at least once a month and urine tests once every 3 months. The local laboratory visits and follow-up visits at the NIH Clinical Center will help the study team determine whether the HPTH treatment is controlling your hypoparathyroidism.

DETAILED DESCRIPTION:
Objectives

The primary objective of this study is to evaluate the skeletal effects of hormone replacement therapy with HPTH in hypoparathyroidism.

Study Population

This study will enroll up to 69 subjects with physician-diagnosed hypoparathyroidism.<TAB>

Design

This study will treat hypoparathyroid individuals with synthetic human PTH 1-34 (HPTH) for up to 5 years, periodically assessing skeletal changes through biochemical markers and iliac-crest bone biopsies, which will allow for ultrastructural, cellular, and molecular analyses.

With respect to HPTH treatment, this study is a single group, within-subjects, repeated measures treatment trial. With respect to all bone biopsy analyses, the design is a parallel group design with each subject allocated to one of the 3 biopsy follow-up times: 1, 2 or 4 years after initiation of HPTH therapy. Post-baseline biopsy timing will be randomly assigned (1:1.2:1.4, respectively) to each subject, stratified by gender and by menopausal status, when relevant. Changes from baseline (time 0) to 1, 2 and 4-years will be compared. Subjects who were on conventional therapy in the former version of the protocol will also be randomized into the new study design. In contrast to new subjects, whose biopsy is performed at the end of the conventional care run-in period, the pre-conventional care biopsy will be used as the baseline for the those subjects entering the new design after having been on conventional care in the older protocol. Because it is not known with certainty what effects duration of time on conventional therapy will have on biopsy results, randomization will also be stratified on status of prior study participation. The subjects who were on HPTH therapy at the time of the protocol redesign are followed as a separate group under this protocol.

Outcome Measures

Primary:

Changes in static and dynamic bone histomorphometry after 1 year, 2 years, and 4 years of HPTH therapy. Primary outcome measurements include:

* Mineralized perimeter
* Bone formation rate
* Cortical width
* Cortical area
* Osteoid width
* Osteoid perimeter
* Mineral apposition rate

Secondary:

Changes in bone mineralization density distribution at 1, 2 and 4 years of HPTH therapy. The specific outcomes that will be measured include:

* Spectral calcium-mean
* Calcium-peak
* Calcium-width

Changes from baseline will be assessed in the following outcomes:

* Biochemical markers of bone metabolism: osteocalcin, bone-specific alkaline phosphatase, collagen cross-linked N-telopeptide.
* Serum and urine calcium; 1,25-OH2-Vitamin D
* Bone density assessed by DXA and quantitative CT
* Nephrocalcinosis by ultrasound and CT
* Fatigue Symptom Inventory
* 6-Minute Walk Test
* SF-36 Health Survey

Tertiary:

Changes in blood chemistries and FGF23, renal mineral handling, and PTH sensitivity with the initiation of HPTH, which include:

* Serum albumin, calcium, phosphorus, magnesium, sodium, potassium, chloride, Total CO2, creatinine, glucose, urea nitrogen, and FGF23
* Urine cAMP, creatinine, phosphorus, calcium, and pH

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age eligibility at screening:

     1. Premenopausal women: aged 18 to 45 years,
     2. Postmenopausal women: aged greater than or equal to 53 years to 70 years and 5 years since last menses. For women without a uterus, subjects must have a clinical history of menopause for at least 5 years and an FSH greater than 30 U/L.
     3. Men: aged 18 to 70 years,
  2. Physician-diagnosed hypoparathyroidism of at least 1-year duration, confirmed by medical record review. The investigators will confirm the diagnosis during the screening visit at which time the subject must have an intact PTH < 30 pg/mL.

EXCLUSION CRITERIA:

1. Moderate to severe hepatic disease defined as hepatic transaminases (ALT and AST) > 2 times the upper limit of normal
2. Severe renal insufficiency defined as a calculated GFR < 25 mL/min/1.73 m(2), using the CKD-EPI equation(15).
3. Allergy or intolerance to tetracycline antibiotics
4. Pregnant or lactating or planning to become pregnant during the course of the study. (Women who are able to get pregnant must agree to use an effective form of birth control while in this study.).
5. Perimenopausal defined by no menses for 6 months to 5 years and an FSH > 20 U/L at the screening and/or baseline visits..
6. Chronic diseases that might affect mineral metabolism such as diabetes, celiac disease, Crohn s disease, Cushing s syndrome, or adrenal insufficiency
7. Concurrent treatment with doses of thyroid hormone intended to suppress thyroid stimulating hormone below the assay s detection limit or persistent thyroid cancer
8. History of a skeletal disease unrelated to hypoparathyroidism, such as osteoporosis or low bone density (defined as a DXA Z-Score < -2 in all subjects or T-score < -2 in subjects greater than or equal to 20 year old), osteosarcoma, Paget s disease, alkaline phosphatase > 1.5 times the upper limit of normal, or metastatic bone disease
9. History of retinoblastoma or Li-Fraumeni syndrome
10. History of treatment with bisphosphonates, calcitonin, tamoxifen, selective-estrogen receptor modulators, or directed skeletal irradiation
11. Use of oral or intravenous corticosteroids or estrogen replacement therapy for more than 3 weeks within the last 6 months
12. Use of depot medroxyprogesterone for contraception within the past 12 months
13. Chronic inadequate biochemical control with conventional therapy and/or calcium infusion dependent
14. Seizure disorder requiring antiepileptic medications
15. Treatment with PTH for more than 2 weeks continuously at any time, prior to study entry
16. Any cognitive impairment that limits the subject s ability to comply, independently or through the assistance of a legally authorized representative, with protocol procedures.
17. Open epiphyses as determined by an X-ray of the hand and wrist in subjects < 21 years of age.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-10-30; Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel I Gafni, M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chan JC, Young RB, Alon U, Mamunes P. Hypercalcemia in children with disorders of calcium and phosphate metabolism during long-term treatment with 1,25-dihydroxyvitamin-D3. Pediatrics. 1983 Aug;72(2):225-33. No abstract available. PMID 6688127
- [Background] Chan JC, Young RB, Hartenberg MA, Chinchilli VM. Calcium and phosphate metabolism in children with idiopathic hypoparathyroidism or pseudohypoparathyroidism: effects of 1,25-dihydroxyvitamin D3. J Pediatr. 1985 Mar;106(3):421-6. doi: 10.1016/s0022-3476(85)80668-5. PMID 3838346
- [Background] Christiansen C, Rodbro P, Christensen MS, Hartnack B, Transbol I. Deterioration of renal function during treatment of chronic renal failure with 1,25-dihydroxycholecalciferol. Lancet. 1978 Sep 30;2(8092 Pt 1):700-3. doi: 10.1016/s0140-6736(78)92702-2. PMID 80633
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-D-0016.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals with hypoparathyroidism were enrolled at the NIH clinical center, beginning in October 2006. The protocol was redesigned and amended in February 2010. Some of the previously enrolled participants were re-enrolled in the new study. New participants were also enrolled on the new study through October 2014.
Pre-assignment Details: All participants were put on conventional care therapy for 2-6 months prior to HPTH therapy. Previously enrolled participants had their baseline bone biopsy prior to the study's conventional care period. Newly enrolled participants had their baseline bone biopsy performed at the started of HPTH therapy.
Groups:
- Cohort 1: Received HPTH on Original Protocol: Treated with HPTH therapy on original protocol
- Cohort 2: Received Conventional Care on Original Protocol: Treated with conventional care (CC) throughout original protocol
- Cohort 3: Newly Enrolled No Prior Participation: New participants in revised protocol
Period: Overall Study
Arm/Group | Cohort 1: Received HPTH on Original Protocol | Cohort 2: Received Conventional Care on Original Protocol | Cohort 3: Newly Enrolled No Prior Participation
Started (Previously enrolled in original protocol or (for Cohort 3) newly enrolled in current protocol) | 8 | 15 | 23
Signed Consent to the New Protocol | 7 | 5 | 23
Received HPTH on New Protocol (This category identifies the subset of subjects in the Safety Population.) | 7 | 5 | 19
Randomized to Bone Biopsy Year 1 | 0 | 1 | 5
Randomized to Bone Biopsy Year 2 | 0 | 2 | 6
Randomized to Bone Biospy Year 4 | 0 | 2 | 8
Completed Bone Biopsy Year 1 | 0 | 1 | 4
Completed Bone Biopsy Year 2 | 0 | 2 | 3
Completed Bone Biopsy Year 4 | 0 | 1 | 1
Completed (Completed 5 years of HPTH therapy and 6 month safety follow-up visit.) | 5 | 2 | 0
Not Completed | 3 | 13 | 23
Not completed — Did not re-consent to revised protocol | 1 | 10 | 0
Not completed — FDA partial hold on PTH | 0 | 0 | 11
Not completed — Failed screening | 0 | 0 | 4
Not completed — Switch to Natpara | 0 | 0 | 3
Not completed — Adverse Event | 1 | 0 | 2
Not completed — DXA or QCT z-score or t-score<-2 | 0 | 2 | 0
Not completed — Non-compliance with study protocol | 0 | 1 | 0
Not completed — PTH resistance | 0 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Partial recovery of parathyroid function | 0 | 0 | 1
Not completed — Participant elected to discontinue | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: The Safety Population will consist of all enrolled subjects (all cohorts) who have started any study treatment including, but not limited to, conventional care. This population will be used for safety data summaries.
Groups:
- Cohort 1 (HPTH on Old Study) and Received HPTH on New Study: Cohort 1 was treated with HPTH therapy on original protocol. Cohort 1 participants who consented to the new protocol and were treated with HPTH on the new protocol were followed for safety outcomes only. The Safety population of Cohort 1 consisted of 7 participants.
- Cohort 2 (CC on Old Study) and Treated With HPTH on New Study: Cohort 2 consists of participants previously treated with conventional care (CC) throughout the original protocol. Cohort 2 participants who received at least one dose of HPTH on the new protocol were included in safety population. Cohort 2 safety population includes 5 participants.
- Cohort 3 (Newly Enrolled) and Treated With HPTH on New Study: Cohort 3 consists of new participants (i.e. not previously enrolled) that consented to the revised protocol. The Cohort 3 safety population includes 19 subjects who received any HPTH on the new study.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (HPTH on Old Study) and Received HPTH on New Study | Cohort 2 (CC on Old Study) and Treated With HPTH on New Study | Cohort 3 (Newly Enrolled) and Treated With HPTH on New Study | Total
Number analyzed (Participants) | 7 | 5 | 19 | 31
Age, Customized [Count of Participants; unit: Participants]
  Age: < 20 years | 2 | 0 | 0 | 2
  Age: 20-29 years | 0 | 0 | 2 | 2
  Age: 30-39 years | 1 | 1 | 6 | 8
  Age: 40-49 years | 3 | 3 | 7 | 13
  Age: 50-59 years | 1 | 1 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 16 | 25
  Male | 1 | 2 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 5 | 19 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 5 | 18 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 72.2 (14.39) | 74.9 (21.92) | 82.6 (19.01) | 79.0 (18.56)
Height [Mean (Standard Deviation); unit: cm] — Population: Baseline height was missing for some participants.
  cm
    number analyzed (Participants) | 3 | 0 | 7 | 10
    (all) | 160.8 (6.93) |  | 171.1 (9.67) | 168.0 (9.89)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Since some participants had missing height measures, the BMI could not be calculated for these participants.
  kg/m^2
    number analyzed (Participants) | 3 | 0 | 7 | 10
    (all) | 29.71 (2.232) |  | 29.14 (6.310) | 29.31 (5.266)

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Biopsy Cancellous Bone Volume (Cn.BV/TV)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, so the 2-, and 4-year biopsies were collapsed into one biopsy year group. Cn.BV/TV is one of 8 primary endpoints measured from the bone biopsy. The changes in Cn.BV/TV outcome between two time-points are being reported. The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes.
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: The Bone Biopsy Analysis Population was used for the primary bone biopsy biomarkers. The Bone Biopsy Population consisted of all participants in Cohorts 2 and 3 who completed both their baseline and randomized 1, 2, or 4 year bone biopsies.
Measure: Least Squares Mean (Standard Error); unit: z-score
Groups:
- Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined: Cohort 2 consists of participants previously treated with conventional care (CC) throughout the original protocol. Cohort 3 consisted of all new participants. Efficacy outcomes were only analyzed for Cohorts 2 and 3. (Cohort 1 consisted of previously enrolled participants who were on HPTH therapy on the original protocol and continued on HPTH on the new study as a separate group. These participants were not randomized to a bone biopsy year, nor did they have additional biopsies performed. Cohort 1 participants were followed for safety outcomes only. )
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 12
z-score
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 5
  Biopsy Year 1 - Baseline | 3.05 (1.095)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 3.69 (0.940)
  Biopsy Years 2 and 4 (combined) - Year 1 | 0.64 (1.379)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Cn.BV/TV at biopsy baseline, year 1, 2 & 4 combined as the dependent variable; biopsy year as the independent variable, covariate for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2. No bone biopsy baseline covariate was included because it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the cn.BV/TV between the baseline and the year 1 biopsy; p = 0.015, Mixed Models Analysis — No adjustments were made for multiple comparisons, since the study was terminated early resulting in only 5, 5, and 2 participants having their biopsies at 1, 2, and 4 years respectively
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Cn.BV/TV at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2. No bone biopsy baseline covariate included because it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the cn.BV/TV between the baseline and the years 2 and 4 (combined) biopsy; p = 0.002, Mixed Models Analysis — No adjustments were made for multiple comparisons, because the study was terminated early resulting in only 5, 5, and 2 participants having their biopsies at 1, 2, and 4 years respectively
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis was performed with: Cn.BV/TV change from baseline at biopsy year 1 or years 2 and 4 combined as the dependent variable; biopsy year, and baseline Cn.BV/TV, as model covariates; and a random effect for participant. Since Cohort 2 had a time delay of 30 to 31 months from the baseline biopsy to start of HPTH therapy, this time delay (centered to stabilize variance) was added as a covariate to the model for Cohort 2 only (using a Cohort 2 indicator variable); Test type: Equivalence — A contrast statement within the mixed models analysis tested for differences in the cn.BV/TV between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.649, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Change in Total Number of Cortical Pores Per mm^2 (Ct.Po.N)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, so the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ct.Po.N is a bone biopsy measure that assess the amount of holes in the cortical bone within a predetermined area of cortical bone. The changes in Cn.BV/TV outcome between two time-points are being reported. Cortical bone with a higher number of holes may be at greater risk of fracture. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cortical pores/mm^2
Groups:
- Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined: Cohort 2 consists of participants previously treated with conventional care (CC) throughout the original protocol. Cohort 3 consisted of all new participants. Efficacy outcomes were only analyzed for Cohorts 2 and 3. (Cohort 1 consisted of previously enrolled participants who were on HPTH therapy on the original protocol and continued on HPTH on the new study as a separate group. These participants were not randomized to a bone biopsy year, nor did they have additional biopsies performed. Cohort 1 participants were followed for safety outcomes only.)
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
cortical pores/mm^2
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 1.12 (1.214)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 1.86 (1.149)
  Biopsy Years 2 and 4 (combined) - Year 1 | 0.74 (1.175)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ct.Po.N at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ct.Po.N between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ct.Po.N values for both their baseline and year 1 biopsies; p = 0.371, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis was performed with: Ct.Po.N change from baseline at biopsy year 1 or years 2 and 4 combined as the dependent variable; biopsy year, and baseline Ct.Po.N, as model covariates; and a random effect for participant. Since Cohort 2 had a time delay of 30 to 31 months from the baseline biopsy to start of HPTH therapy, this time delay (centered to stabilize variance) was added as a covariate to the model for Cohort 2 only (using a Cohort 2 indicator variable); Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ct.Po.N between the baseline and the years 2 and 4 (combined) biopsy; p = 0.129, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — A contrast statement within the mixed models analysis tested for differences in the Ct.Po.N between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.538, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Change in Cancellous Bone Formation Rate Per Unit of Bone Surface (Cn.BFR/BS)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Cn.BFR/BS, measured from the bone biopsy, is the cancellous bone formation rate per unit of bone surface where cancellous refers to the spongy structure of the bone. The changes in Cn.BFR/BS between two time-points are being reported. The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes.
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 12
z-score
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 5
  Biopsy Year 1 - Baseline | 4.25 (1.420)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 5.75 (1.251)
  Biopsy Years 2 and 4 (combined) - Year 1 | 1.50 (1.647)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Cn.BFR/BS at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.BFR/BS between the baseline and the year 1 biopsy; p = 0.009, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; A baseline covariate not added to model since it would over-parameterize the model
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 3, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.BFR/BS between the baseline and the years 2 and 4 (combined) biopsy; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — A contrast statement within the mixed models analysis tested for differences in the Cn.BFR/BS between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.374, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

4. Primary Outcome: Change in Cancellous Mineralizing Surface (Bone Surface Based)(Cn.MS/BS)
Description: Following their baseline bone biopsy, 5, 5, and 2 participants were randomized to receive their second bone biopsy at years 1, 2, and 4 after the start of HPTH therapy, respectively. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced in size due to withdrawal and the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Cn.MS/BS is measured from the bone biopsy. This measure demonstrates the percentage of the cancellous bone surface that is actively forming bone. The region of interest is the predefined area of total bone that is being measured. The changes in Cn.MS/BS between two time-points are being reported.
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of predefined area of bone
Groups:
- Cohorts 2 and 3 Combined: Cohort 1 consisted of previously enrolled participants who were on HPTH therapy, were re-consented, and allowed to continue on the current study as a separate group. These participants were not randomized to a bone biopsy year, nor did they have additional biopsies performed. Cohort 1 participants were followed for safety outcomes only. Cohort 2 were previously enrolled participants on conventional care, were re-consented, re-enrolled, and randomized to a biopsy year. Cohort 3 consisted of all new participants consent, enrolled and randomized to a biopsy year. Efficacy outcomes were only analyzed for Cohorts 2 and 3 combined.
Arm/Group | Cohorts 2 and 3 Combined
Number analyzed (Participants) | 12
percentage of predefined area of bone
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 5
  Biopsy Year 1 - Baseline | 14.63 (3.996)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 21.47 (3.489)
  Biopsy Years 2 and 4 (combined) - Year 1 | 6.85 (4.774)
Statistical Analysis 1: Comparison: Cohorts 2 and 3 Combined; Mixed models analysis: Cn.MS/BS at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.MS/BS between the baseline and the year 1 biopsy; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 and 3 Combined; [analysis description as in outcome 4, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.MS/BS between the baseline and the years 2 and 4 (combined) biopsy; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 and 3 Combined; [analysis description as in outcome 4, analysis 1]; Test type: Equivalence — A contrast statement within the mixed models analysis tested for differences in the Cn.MS/BS between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.168, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

5. Primary Outcome: Change in Endocortical Bone Formation Rate Per Unit of Bone Surface (Ec.BFR/BS)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. However, because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ec.BFR/BS is measured from the bone biopsy. This measures the rate of new bone formation per day on the inner cortical (endocortical) surface in a predefined region of cortical bone. The changes in Ec.BFR/BS between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: um^2/um/d
Groups:
- Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. The randomization to a biopsy year provided the opportunity to compare the effects of PTH across-time, in a cross-sectional manner. However, because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group.
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
um^2/um/d
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 0.12 (0.063)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 0.22 (0.055)
  Biopsy Years 2 and 4 (combined) - Year 1 | 0.10 (0.072)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ec.BFR/BS at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.BFR/BS between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ec.BFR/BS values for both their baseline and year 1 biopsies; p = 0.083, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 5, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.BFR/BS between the baseline and the years 2 and 4 (combined) biopsy; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 5, analysis 1]; Test type: Equivalence — A contrast statement within the mixed models analysis tested for differences in the Ec.BFR/BS between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.164, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

6. Primary Outcome: Change in Endocortical Mineralizing Surface (Bone Surface Based) (Ec.MS/BS)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ec.MS/BS is measured from the bone biopsy. This measure demonstrates the percentage of the endocortical bone surface that is actively forming bone. The region of interest is the predefined area of total bone that is being measured. The changes in Ec.MS/BS between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: The Bone Biopsy Analysis Population was used for the primary bone biopsy biomarkers. The Bone Biopsy Population consisted of all participants who completed both their baseline and randomized 1, 2, or 4 year bone biopsies. This will only include participants from cohorts 2 and 3.
Measure: Least Squares Mean (Standard Error); unit: percentage of regional interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
percentage of regional interest
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 18.39 (7.748)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 30.94 (6.757)
  Biopsy Years 2 and 4 (combined) - Year 1 | 12.55 (8.944)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ec.MS/BS at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.MS/BS between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ec.MS/BS values for both their baseline and year 1 biopsies; p = 0.031, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 6, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.MS/BS between the baseline and the years 2 and 4 (combined) biopsy; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 6, analysis 1]; Test type: Equivalence — A contrast statement within the mixed models analysis tested for differences in the Ec.MS/BS between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.178, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

7. Primary Outcome: Change in Intracortical Bone Formation Rate Per Unit of Bone Surface (Ic.BFR/BS)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. However, because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ic.BFR/BS is measured from the bone biopsy. This measures the rate of new bone formation between the two cortical surfaces (intracortical) in a predefined region of cortical bone. The changes in Ic.BFR/BS between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: um^2/um/d
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
um^2/um/d
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 0.18 (0.045)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 0.10 (0.040)
  Biopsy Years 2 and 4 (combined) - Year 1 | -0.07 (0.052)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ic.BFR/BS at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.BFR/BS between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ic.BFR/BS values for both their baseline and year 1 biopsies; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 7, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.BFR/BS between the baseline and the years 2 and 4 (combined) biopsy; p = 0.022, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 7, analysis 1]; Test type: Equivalence — A contrast statement within the mixed models analysis tested for differences in the Ic.BFR/BS between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.172, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

8. Primary Outcome: Change in Intracortical Mineralizing Surface (Bone Surface Based) (Ic.MS/BS)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ic.MS/BS is measured from the bone biopsy. This measure demonstrates the percentage of the intracortical bone surface that is actively forming bone. The region of interest is the predefined area of total bone that is being measured. The changes in Ic.MS/BS between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of regional interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
percentage of regional interest
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 24.75 (6.000)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 14.36 (5.208)
  Biopsy Years 2 and 4 (combined) - Year 1 | -10.4 (6.999)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ic.MS/BS at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.MS/BS between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ic.MS/BS values for both their baseline and year 1 biopsies; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 8, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.MS/BS between the baseline and the years 2 and 4 (combined) biopsy; p = 0.018, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 8, analysis 1]; Test type: Equivalence — A contrast statement within the mixed models analysis tested for differences in the Ic.MS/BS between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.155, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change in Trabecular Thickness (Tb.Th)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Tb.Th is measured from the bone biopsy. Tb.Th is the mean thickness of trabeculae, assessed using direct 3D methods. The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes. The changes in Tb.Th between two time-points are being reported.
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 12
z-score
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 5
  Biopsy Year 1 - Baseline | -0.28 (0.779)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 0.05 (0.675)
  Biopsy Years 2 and 4 (combined) - Year 1 | 0.33 (0.950)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Tb.Th at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Tb.Th between the baseline and the year 1 biopsy; p = 0.720, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 9, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Tb.Th between the baseline and the years 2 and 4 (combined) biopsy; p = 0.944, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 9, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Tb.Th between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.730, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change in Trabecular Number (Tb.N)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Tb.N is measured from the bone biopsy. Tb.N is the measure of the average number of trabeculae per unit length. The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes. The changes in Tb.N between two time-points are being reported.
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 12
z-score
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 5
  Biopsy Year 1 - Baseline | 3.62 (1.382)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 3.30 (1.221)
  Biopsy Years 2 and 4 (combined) - Year 1 | -0.32 (1.586)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis was performed with: Tb.N change from baseline at biopsy year 1 or years 2 and 4 combined as the dependent variable; biopsy year, and baseline Tb.N, as model covariates; and a random effect for participant. Since Cohort 2 had a time delay of 30 to 31 months from the baseline biopsy to start of HPTH therapy, this time delay (centered to stabilize variance) was added as a covariate to the model for Cohort 2 only (using a Cohort 2 indicator variable); Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Tb.N between the baseline and the year 1 biopsy; p = 0.019, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 10, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Tb.N between the baseline and the years 2 and 4 (combined) biopsy; p = 0.017, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 10, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Tb.N between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.843, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Change in Trabecular Separation (Tb.Sp)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Tb.Sp is measured from the bone biopsy. Tb.Sp is the mean distance between trabeculae, assessed using direct 3D methods. The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes. The changes in Tb.Sp between two time-points are being reported.
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 12
z-score
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 5
  Biopsy Year 1 - Baseline | -2.28 (0.803)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | -1.76 (0.693)
  Biopsy Years 2 and 4 (combined) - Year 1 | 0.52 (0.997)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Tb.Sp at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Tb.Sp between the baseline and the year 1 biopsy; p = 0.013, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 11, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Tb.Sp between the baseline and the years 2 and 4 (combined) biopsy; p = 0.025, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 11, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Tb.Sp between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.608, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

12. Secondary Outcome: Change in Average Thickness of Inner and Outer Cortices (Ct.Th)
Description: Participants (Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ct.Th, measured from the bone biopsy, is the average thickness of the inner and outer cortices. The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes. The changes in Ct.Th between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
z-score
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 2.02 (0.916)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 0.78 (0.771)
  Biopsy Years 2 and 4 (combined) - Year 1 | -1.25 (1.092)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ct.Th at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ct.Th between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ct.Th values for both their baseline and year 1 biopsies; p = 0.043, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 12, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ct.Th between the baseline and the years 2 and 4 (combined) biopsy; p = 0.334, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis was performed with: Ct.Th change from baseline at biopsy year 1 or years 2 and 4 combined as the dependent variable; biopsy year, and baseline Ct.Th, as model covariates; and a random effect for participant. Since Cohort 2 had a time delay of 30 to 31 months from the baseline biopsy to start of HPTH therapy, this time delay (centered to stabilize variance) was added as a covariate to the model for Cohort 2 only (using a Cohort 2 indicator variable); Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ct.Th between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.269, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

13. Secondary Outcome: Total Area of Inner and Outer Cortices (Ct.Ar)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ct.AR is measured from the bone biopsy. This measure defines the area of the outer cortex and inner cortex within a predefined section of cortical bone. The changes in Ct.Ar between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of region of interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
percentage of region of interest
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 6.56 (6.905)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 1.93 (6.128)
  Biopsy Years 2 and 4 (combined) - Year 1 | -4.64 (8.006)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ct.Ar at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ct.Ar between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ct.Ar values for both their baseline and year 1 biopsies; p = 0.358, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 13, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ct.Ar between the baseline and the years 2 and 4 (combined) biopsy; p = 0.760, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 13, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ct.Ar between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.570, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

14. Secondary Outcome: Change in Total Area of Cortical Porosity (Ct.Po.Ar)
Description: Following their baseline bone biopsy, 5, 5, and 2 participants were randomized to receive their second bone biopsy at years 1, 2, and 4 after the start of HPTH therapy, respectively. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced in size due to withdrawal and the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ct.Po.Ar is measured from the bone biopsy. This measure defines the area of the cortical bone with holes within a predefined section of cortical bone. The changes in Tb.Sp between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percentage of region of interest
Arm/Group | Cohorts 2 and 3 Combined
Number analyzed (Participants) | 11
percentage of region of interest
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 3.41 (2.337)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 0.26 (1.911)
  Biopsy Years 2 and 4 (combined) - Year 1 | -3.15 (2.837)
Statistical Analysis 1: Comparison: Cohorts 2 and 3 Combined; Mixed models analysis: Ct.Po.Ar at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ct.Po.Ar between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ct.Po.Ar values for both their baseline and year 1 biopsies; p = 0.166, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 and 3 Combined; [analysis description as in outcome 14, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ct.Po.Ar between the baseline and the years 2 and 4 (combined) biopsy; p = 0.895, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 and 3 Combined; [analysis description as in outcome 14, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ct.Po.Ar between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.282, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

15. Secondary Outcome: Change in Cancellous Osteoid Thickness (Cn.O.Th)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Cn.O.Th measured from the bone biopsy. This measures the thickness of the unmineralized bone (osteoid) in a predefined region of cancellous bone. The changes in Cn.O.Th between two time-points are being reported.
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: um
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 12
um
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 5
  Biopsy Year 1 - Baseline | 1.99 (0.553)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 2.29 (0.472)
  Biopsy Years 2 and 4 (combined) - Year 1 | 0.30 (0.704)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Cn.O.Th at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.O.Th between the baseline and the year 1 biopsy; p = 0.003, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 15, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.O.Th between the baseline and the years 2 and 4 (combined) biopsy; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 15, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.O.Th between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.680, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

16. Secondary Outcome: Change in Cancellous Bone Mineral Apposition Rate (Cn.MAR)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Cn.MAR is measured from the bone biopsy. This measures the rate mineral is being laid down per day in a predefined region of the cancellous bone. The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes. The changes in Cn.MAR between two time-points are being reported.
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 12
z-score
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 5
  Biopsy Year 1 - Baseline | 3.21 (1.002)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 3.07 (0.885)
  Biopsy Years 2 and 4 (combined) - Year 1 | -0.14 (1.151)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Cn.MAR at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.MAR between the baseline and the year 1 biopsy; p = 0.006, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 16, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.MAR between the baseline and the years 2 and 4 (combined) biopsy; p = 0.004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 16, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.MAR between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.904, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

17. Secondary Outcome: Change in Cancellous Osteoid Surface / Bone Surface (Cn.OS/BS)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Cn.OS/BS is measured from the bone biopsy. This measure demonstrates the percentage of the cancellous bone surface that contains unmineralized bone (osteoid). The region of interest is the predefined area of total bone that is being measured. The changes in Cn.OS/BS between two time-points are being reported.
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of region of interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 12
percentage of region of interest
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 5
  Biopsy Year 1 - Baseline | 12.70 (3.407)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 24.34 (2.971)
  Biopsy Years 2 and 4 (combined) - Year 1 | 11.64 (4.084)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Cn.OS/BS at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.OS/BS between the baseline and the year 1 biopsy; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 17, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.OS/BS between the baseline and the years 2 and 4 (combined) biopsy; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 17, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.OS/BS between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.010, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

18. Secondary Outcome: Change in Cancellous Eroded Surface / Bone Surface (Cn.ES/BS)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Cn.ES/BS is measured from the bone biopsy. This measure demonstrates the percentage of the cancellous bone surface that contains unmineralized bone (osteoid). The region of interest is the predefined area of total bone that is being measured. The changes in Cn.ES/BS between two time-points are being reported.
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of region of interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 12
percentage of region of interest
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 5
  Biopsy Year 1 - Baseline | 6.55 (1.648)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 10.30 (1.543)
  Biopsy Years 2 and 4 (combined) - Year 1 | 3.75 (1.415)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Cn.ES/BS at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.ES/BS between the baseline and the year 1 biopsy; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 18, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.ES/BS between the baseline and the years 2 and 4 (combined) biopsy; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 18, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.ES/BS between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.020, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

19. Secondary Outcome: Change in Cancellous Adjusted Apposition Rate (Cn.AjAR)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Cn.AjAR is measured from the bone biopsy. Cn.AjAR represents the Cn.MAR averaged over the entire osteoid surface.The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes. The changes in Cn.AjAR between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
z-score
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 5
  Biopsy Year 1 - Baseline | 3.10 (0.824)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 6
  Biopsy Years 2 and 4 (combined) - Baseline | 1.89 (0.722)
  Biopsy Years 2 and 4 (combined) - Year 1 | -1.21 (0.972)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Cn.AjAR at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.AjAR between the baseline and the year 1 biopsy; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 19, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.AjAR between the baseline and the years 2 and 4 (combined) biopsy; p = 0.022, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 19, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cn.AjAR between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.228, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

20. Secondary Outcome: Change in Endocortical Osteoid Thickness (Ec.O.Th)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ec.O.Th is measured from the bone biopsy. This measures the thickness of the unmineralized bone (osteoid) on the inner side of the cortex(endocortical). The changes in Cn.AjAR between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: um
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
um
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 2.15 (0.628)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 1.84 (0.552)
  Biopsy Years 2 and 4 (combined) - Year 1 | -0.31 (0.718)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ec.O.Th at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.O.Th between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ec.O.Th values for both their baseline and year 1 biopsies; p = 0.004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 20, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.O.Th between the baseline and the years 2 and 4 (combined) biopsy; p = 0.006, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 20, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.O.Th between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.670, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

21. Secondary Outcome: Change in Endocortical Bone Mineral Apposition Rate (Ec.MAR)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose.Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ec.MAR is measured from the bone biopsy. This measures the rate mineral is being laid down per day on the inner cortical (endocortical) surface in a predefined region of cortical bone. The changes in Ec.MAR between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: um/d
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
um/d
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 0.41 (0.115)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 0.46 (0.104)
  Biopsy Years 2 and 4 (combined) - Year 1 | 0.05 (0.126)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ec.MAR at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.MAR between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ec.MAR values for both their baseline and year 1 biopsies; p = 0.003, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 21, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.MAR between the baseline and the years 2 and 4 (combined) biopsy; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 21, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.MAR between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.712, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

22. Secondary Outcome: Change in Endocortical Osteoid Surface / Bone Surface (Ec.OS/BS)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ec.OS/BS is measured from the bone biopsy. This measures the rate mineral is being laid down per day on the inner cortical (endocortical) surface in a predefined region of cortical bone. The changes in Ec.OS/BS between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of region of interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
percentage of region of interest
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 13.43 (5.606)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 24.56 (4.872)
  Biopsy Years 2 and 4 (combined) - Year 1 | 11.13 (6.491)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ec.OS/BS at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.OS/BS between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ec.OS/BS values for both their baseline and year 1 biopsies; p = 0.029, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 22, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.OS/BS between the baseline and the years 2 and 4 (combined) biopsy; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 22, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.OS/BS between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.104, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

23. Secondary Outcome: Change in Endocortical Eroded Surface / Bone Surface (Ec.ES/BS)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4- year biopsies were collapsed into one biopsy year group. Ec.ES/BS is measured from the bone biopsy. This measure demonstrates the percentage of the endocortical bone surface that is resorbed (eroded). The region of interest is the predefined area of total bone that is being measured. The changes in Ec.ES/BS between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of region of interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
percentage of region of interest
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 5.95 (3.270)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 9.29 (3.063)
  Biopsy Years 2 and 4 (combined) - Year 1 | 3.34 (3.288)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ec.ES/BS at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.ES/BS between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ec.ES/BS values for both their baseline and year 1 biopsies; p = 0.088, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 23, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.ES/BS between the baseline and the years 2 and 4 (combined) biopsy; p = 0.009, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 23, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.ES/BS between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.325, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

24. Secondary Outcome: Change in Endocortical Adjusted Apposition Rate (Ec.AjAR)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ec.AjAR is measured from the bone biopsy. Ec.AjAR represents the endocortical mineral apposition rate (Ec.MAR) averaged over the entire osteoid surface. This is another histomorphometric way to evaluate the rate at which bone is laid down on the inner cortical surface per day. The changes in Ec.AjAR between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: um/d
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 8
um/d
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 3
  Biopsy Year 1 - Baseline | 0.50 (0.109)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 5
  Biopsy Years 2 and 4 (combined) - Baseline | 0.49 (0.088)
  Biopsy Years 2 and 4 (combined) - Year 1 | -0.00 (0.135)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ec.AjAR at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.AjAR between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 3 participants with non-missing Ec.AjAR values for both their baseline and year 1 biopsies; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 24, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.AjAR between the baseline and the years 2 and 4 (combined) biopsy; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 24, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ec.AjAR between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.974, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

25. Secondary Outcome: Change in Intracortical Osteoid Thickness (Ic.O.Th)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ic.O.Th is one of 21 secondary endpoints measured from the bone biopsy. This measures the thickness of the unmineralized bone (osteoid) within the middle of the cortex (intracortical). The changes in Ic.O.Th between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: um
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
um
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 2.39 (0.687)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 1.48 (0.564)
  Biopsy Years 2 and 4 (combined) - Year 1 | -0.91 (0.833)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ic.O.Th at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.O.Th between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ic.O.Th values for both their baseline and year 1 biopsies; p = 0.004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 25, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.O.Th between the baseline and the years 2 and 4 (combined) biopsy; p = 0.023, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 25, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.O.Th between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.288, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

26. Secondary Outcome: Change in Intracortical Bone Mineral Apposition Rate (Ic.MAR)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ic.MAR is measured from the bone biopsy. This measures the rate mineral is being laid down per day within the middle of the cortex (intracortical) surface in a predefined region of cortical bone. The changes in Ic.MAR between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: um/d
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
um/d
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 0.23 (0.174)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 0.12 (0.161)
  Biopsy Years 2 and 4 (combined) - Year 1 | -0.12 (0.185)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ic.MAR at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.MAR between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ic.MAR values for both their baseline and year 1 biopsies; p = 0.202, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 26, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.MAR between the baseline and the years 2 and 4 (combined) biopsy; p = 0.486, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 26, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.MAR between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.535, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

27. Secondary Outcome: Change in Intracortical Osteoid Surface / Bone Surface (Ic.OS/BS)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ic.OS/BS measured from the bone biopsy. This measure demonstrates the percentage of the intracortical bone surface that is not mineralized (osteoid). The region of interest is the predefined area of total bone that is being measured. The changes in OS/BS between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of region of interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
percentage of region of interest
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 18.39 (4.284)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 13.17 (3.540)
  Years 2 and 4 (combined) - Year 1 Biopsy | -5.22 (5.181)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ic.OS/BS at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.OS/BS between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ic.OS/BS values for both their baseline and year 1 biopsies; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 27, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.OS/BS between the baseline and the years 2 and 4 (combined) biopsy; p = 0.003, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 27, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.OS/BS between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.328, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

28. Secondary Outcome: Change in Intracortical Eroded Surface / Bone Surface (Ic.ES/BS)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ic.ES/BS is measured from the bone biopsy. This measure demonstrates the percentage of bone surface within the middle of the cortex that is resorbed (eroded). The region of interest is the predefined area of total bone that is being measured. The changes in Ic.ES/BS between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of region of interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
percentage of region of interest
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 6.79 (1.840)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 7
  Biopsy Years 2 and 4 (combined) - Baseline | 7.40 (1.500)
  Biopsy Years 2 and 4 (combined) - Year 1 | 0.61 (2.239)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ic.ES/BS at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.ES/BS between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ic.ES/BS values for both their baseline and year 1 biopsies; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 28, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.ES/BS between the baseline and the years 2 and 4 (combined) biopsy; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 28, analysis 1]; Test type: Equivalence — A contrast statement within the mixed models analysis tested for differences in the Ic.ES/BS between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.789, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

29. Secondary Outcome: Change in Intracortical Adjusted Apposition Rate (Ic.AjAR)
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. Ic.AjAR is one of 21 secondary endpoints measured from the bone biopsy. Ic.AjAR represents the intracortical mineral apposition rate (Ic.MAR) averaged over the the entire osteoid surface. This is another histomorphometric way to evaluate the rate at which bone is laid down within the middle of the cortex per day. The changes in Ic.AjAR between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline values)
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: um/d
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 10
um/d
  Biopsy Year 1 - Baseline: number analyzed (Participants) | 4
  Biopsy Year 1 - Baseline | 0.16 (0.349)
  Biopsy Years 2 and 4 (combined) - Baseline: number analyzed (Participants) | 6
  Biopsy Years 2 and 4 (combined) - Baseline | -0.18 (0.318)
  Biopsy Years 2 and 4 (combined) - Year 1 | -0.34 (0.345)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis: Ic.AjAR at biopsy baseline, year 1, and years 2 and 4 combined as the dependent variable; biopsy year as the independent variable, model covariates for Cohort; and a random effect for participant. Since Cohort 2 had a time delay from the baseline biopsy to start of HPTH therapy, this time delay (centered) was added as a covariate for Cohort 2 (using a Cohort 2 indicator variable). No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.AjAR between the baseline and the year 1 biopsy. P-value interpretation is questionable since there were only 4 participants with non-missing Ic.AjAR values for both their baseline and year 1 biopsies; p = 0.651, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 29, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.AjAR between the baseline and the years 2 and 4 (combined) biopsy; p = 0.580, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 29, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Ic.AjAR between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.338, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

30. Secondary Outcome: Change in Cortex 1 Spectral Calcium Mean From the Back-Scattered Electron Imaging of Bone-Biopsies
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. The Cortex 1 Spectral Calcium Mean is a measure of mean bone calcium content of the bone cortex 1 based on the mineralization density distribution (BMDD) from the back-scattered electron imaging scan of the bone biopsies. The changes in Ic.MAR between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of the region of interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
Percentage of the region of interest
  Year 1 - Baseline Biopsy: number analyzed (Participants) | 5
  Year 1 - Baseline Biopsy | -0.98 (0.357)
  Years 2 and 4 (combined) - Baseline Biopsy: number analyzed (Participants) | 6
  Years 2 and 4 (combined) - Baseline Biopsy | -1.15 (0.633)
  Years 2 and 4 (combined) - Year 1 Biopsy | -0.16 (0.525)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis was performed with Cortex 1 Spectral Calcium Mean as the dependent variable; biopsy year (baseline, year 1, and years 2 and 4 combined) as the independent variable; study cohort as a covariate; and a random effect for participant. No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium Mean between the baseline and the year 1 biopsy; p = 0.020, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 30, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium Mean between the baseline and the years 2 and 4 (combined) biopsy; p = 0.110, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 30, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium Mean between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.764, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

31. Secondary Outcome: Change in Cortex 1 Spectral Calcium Peak From the Back-Scattered Electron Imaging of Bone-Biopsies
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. The Cortex 1 Spectral Calcium Peak is a measure of the most frequent calcium content of the bone cortex 1 based on the bone mineralization density distribution (BMDD) from the back-scattered electron imaging scan of the bone biopsies. The changes in Ic.MAR between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of the region of interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
Percentage of the region of interest
  Year 1 Biopsy - Baseline Biopsy: number analyzed (Participants) | 5
  Year 1 Biopsy - Baseline Biopsy | -0.47 (0.365)
  Years 2 and 4 (combined) - Baseline Biopsy: number analyzed (Participants) | 6
  Years 2 and 4 (combined) - Baseline Biopsy | -0.96 (0.673)
  Years 2 and 4 (combined) - Year 1 Biopsy | -0.49 (0.588)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis was performed with Cortex 1 Spectral Calcium Peak as the dependent variable; biopsy year (baseline, year 1, and years 2 and 4 combined) as the independent variable; study cohort as a covariate; and a random effect for participant. No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium Peak between the baseline and the year 1 biopsy; p = 0.227, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 31, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium Peak between the baseline and the years 2 and 4 (combined) biopsy; p = 0.194, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 31, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium Peak between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.434, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

32. Secondary Outcome: Change in Cortex 1 Spectral Calcium Width From the Back-Scattered Electron Imaging of Bone-Biopsies
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. The Cortex 1 Spectral Calcium Low is a measure of the area of low bone cortex 1 mineralization based on the mineralization density distribution (BMDD) from the back-scattered electron imaging scan of the bone biopsies. The changes in Ic.MAR between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of the region of interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
Percentage of the region of interest
  Year 1 - Baseline Biopsy: number analyzed (Participants) | 5
  Year 1 - Baseline Biopsy | 1.24 (0.343)
  Years 2 and 4 (combined) - Baseline Biopsy: number analyzed (Participants) | 6
  Years 2 and 4 (combined) - Baseline Biopsy | 1.13 (0.302)
  Years 2 and 4 (combined) - Year 1 Biopsy | -0.11 (0.415)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis was performed with Cortex 1 Spectral Calcium Width as the dependent variable; biopsy year (baseline, year 1, and years 2 and 4 combined) as the independent variable; study cohort as a covariate; and a random effect for participant. No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium Width between the baseline and the year 1 biopsy; p = 0.003, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 32, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium Width between the baseline and the years 2 and 4 (combined) biopsy; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 32, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium Width between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.787, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

33. Secondary Outcome: Change in Cortex 1 Spectral Calcium Low From the Back-Scattered Electron Imaging of Bone-Biopsies
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. The Cortex 1 Spectral Calcium Low is a measure of the area of low bone cortex 1 mineralization based on the mineralization density distribution (BMDD) from the back-scattered electron imaging scan of the bone biopsies. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of the region of interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
Percentage of the region of interest
  Year 1 - Baseline Biopsy: number analyzed (Participants) | 5
  Year 1 - Baseline Biopsy | 4.95 (2.172)
  Years 2 and 4 (combined) - Baseline Biopsy: number analyzed (Participants) | 6
  Years 2 and 4 (combined) - Baseline Biopsy | 7.51 (3.245)
  Years 2 and 4 (combined) - Year 1 Biopsy | 2.55 (4.088)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis was performed with Cortex 1 Spectral Calcium Low as the dependent variable; biopsy year (baseline, year 1, and years 2 and 4 combined) as the independent variable; study cohort as a covariate; and a random effect for participant. No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium Low between the baseline and the year 1 biopsy; p = 0.082, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 33, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium Low between the baseline and the years 2 and 4 (combined) biopsy; p = 0.057, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 33, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium Low between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.547, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

34. Secondary Outcome: Change in Cortex 1 Spectral Calcium High From the Back-Scattered Electron Imaging of Bone-Biopsies
Description: Participants (in Cohorts 2 and 3) were randomized to receive their second bone biopsy at year 1, 2, or 4 after the start of HPTH therapy. For Cohort 2, the baseline bone biopsy was completed at the start of CC on the original protocol. For Cohort 3, the baseline biopsy was completed immediately prior to the first HPTH dose. Because the sample sizes for the 1-, 2- and 4-year biopsies are reduced due to the early termination of the study, the 2-, and 4-year biopsies were collapsed into one biopsy year group. The Cortex 1 Spectral Calcium High is a measure of the area of high bone cortex 1 mineralization based on the mineralization density distribution (BMDD) from the back-scattered electron imaging scan of the bone biopsies. The changes in Ic.MAR between two time-points are being reported. The n's in the outcome measure table refer to the number of complete records (non-missing baseline and post-baseline measures).
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of the region of interest
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 11
Percentage of the region of interest
  Year 1 - Baseline Biopsy: number analyzed (Participants) | 5
  Year 1 - Baseline Biopsy | -0.40 (4.052)
  Years 2 and 4 (combined) - Baseline Biopsy: number analyzed (Participants) | 6
  Years 2 and 4 (combined) - Baseline Biopsy | -3.54 (3.592)
  Years 2 and 4 (combined) - Year 1 Biopsy | -3.14 (4.049)
Statistical Analysis 1: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; Mixed models analysis was performed with Cortex 1 Spectral Calcium High as the dependent variable; biopsy year (baseline, year 1, and years 2 and 4 combined) as the independent variable; study cohort as a covariate; and a random effect for participant. No bone biopsy baseline covariate included since it would over-parameterize the model; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium High between the baseline and the year 1 biopsy; p = 0.922, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 34, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium High between the year 1 and the years 2 and 4 (combined) biopsy; p = 0.342, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined; [analysis description as in outcome 34, analysis 1]; Test type: Other — A contrast statement within the mixed models analysis tested for differences in the Cortex 1 Spectral Calcium High between the year 1 biopsy and the years 2 and 4 (combined) biopsy; p = 0.449, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

35. Secondary Outcome: Raw 1/3 Radius Bone Mineralization Density (BMD) Assessed by DXA.
Description: The DXA BMD measures were assessed every 6 months over 5 years, and at a follow-up visit post-HPTH therapy. Due to varying lengths of time on each participant was on HPTH, these BMD assessment times were collapsed for purposes of analysis to: baseline, 6-month on HPTH therapy, last visit on HPTH therapy, and the post-HPTH follow-up visit The 1/3 Radius BMD is one of 6 bone regions measurements of bone mineralization density assessed by DXA.
Time Frame: Baseline, 6-months after start of HPTH, last visit on HPTH (up to 5 years), and post-HPTH follow-up visit (6 months post last visit on HPTH)
Population: Secondary Efficacy Population: This population consists of all participants who received at least one dose of HPTH and had at least one post-baseline non-biopsy efficacy assessment. This population will only include participants in Cohorts 2 and 3.
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
g/cm^2
  Raw BMD at Baseline | 0.746 (0.0138)
  Raw BMD at 6 months | 0.741 (0.0149)
  Raw BMD at last HPTH visit: number analyzed (Participants) | 17
  Raw BMD at last HPTH visit | 0.731 (0.0258)
  Raw BMD at Follow-up: number analyzed (Participants) | 18
  Raw BMD at Follow-up | 0.716 (0.0181)

36. Secondary Outcome: Raw AP Spine Bone Mineralization Density (BMD) Assessed by DXA
Description: The DXA BMD were assessed every 6 months over 5 years, and at a follow-up visit post-HPTH therapy. Due to varying lengths of time on each participant was on HPTH, these BMD assessment times were collapsed for purposes of analysis to: baseline, 6-month on HPTH therapy, last visit on HPTH therapy, and the post-HPTH follow-up visit. The AP Spine BMD is one of 6 bone regions measurements of bone mineralization density assessed by DXA.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
g/cm^2
  Raw BMD at Baseline | 1.175 (0.0253)
  Raw BMD at 6 months | 1.139 (0.0228)
  Raw BMD at last HPTH visit: number analyzed (Participants) | 17
  Raw BMD at last HPTH visit | 1.178 (0.0427)
  Raw BMD at Follow-up: number analyzed (Participants) | 18
  Raw BMD at Follow-up | 1.250 (0.0362)

37. Secondary Outcome: Raw Femoral Neck Bone Mineralization Density (BMD) Assessed by DXA
Description: The DXA BMD measures were assessed every 6 months over 5 years, and at a follow-up visit post-HPTH therapy. Due to varying lengths of time on each participant was on HPTH, these BMD assessment times were collapsed for purposes of analysis to: baseline, 6-month on HPTH therapy, last visit on HPTH therapy, and the post-HPTH follow-up visit. The Femoral BMD is one of 6 bone regions measurements of bone mineralization density assessed by DXA.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
g/cm^2
  Raw BMD at Baseline | 0.909 (0.0234)
  Raw BMD at 6 months | 0.881 (0.0233)
  Raw BMD at last HPTH visit: number analyzed (Participants) | 17
  Raw BMD at last HPTH visit | 0.935 (0.0328)
  Raw BMD at Follow-up: number analyzed (Participants) | 18
  Raw BMD at Follow-up | 0.925 (0.0339)

38. Secondary Outcome: Raw Lateral Spine Bone Mineralization Density (BMD) Assessed by DXA
Description: The DXA BMD were assessed every 6 months over 5 years, and at a follow-up visit post-HPTH therapy. Due to varying lengths of time on each participant was on HPTH, these BMD assessment times were collapsed for purposes of analysis to: baseline, 6-month on HPTH therapy, last visit on HPTH therapy, and the post-HPTH follow-up visit. The Lateral Spine BMD is one of 6 bone regions measurements of bone mineralization density assessed by DXA .
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
g/cm^2
  Raw BMD at Baseline: number analyzed (Participants) | 18
  Raw BMD at Baseline | 0.916 (0.0179)
  Raw BMD at 6 months: number analyzed (Participants) | 18
  Raw BMD at 6 months | 0.918 (0.0215)
  Raw BMD at last HPTH visit: number analyzed (Participants) | 14
  Raw BMD at last HPTH visit | 1.032 (0.0404)
  Raw BMD at Follow-up: number analyzed (Participants) | 13
  Raw BMD at Follow-up | 1.094 (0.0676)

39. Secondary Outcome: Raw Total Hip Bone Mineralization Density (BMD) Assessed by DXA
Description: The DXA BMD measures were assessed every 6 months over 5 years, and at a follow-up visit post-HPTH therapy. Due to varying lengths of time on each participant was on HPTH, these BMD assessment times were collapsed for purposes of analysis to: baseline, 6-month on HPTH therapy, last visit on HPTH therapy, and the post-HPTH follow-up visit. The Total Hip BMD is one of 6 bone regions measurements of bone mineralization density assessed by DXA.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
g/cm^2
  Raw BMD at Baseline | 1.043 (0.0246)
  Raw BMD at 6 months | 1.010 (0.0238)
  Raw BMD at last HPTH visit: number analyzed (Participants) | 17
  Raw BMD at last HPTH visit | 1.043 (0.0301)
  Raw BMD at Follow-up: number analyzed (Participants) | 18
  Raw BMD at Follow-up | 1.045 (0.0279)

40. Secondary Outcome: Raw Whole Body Bone Mineralization Density (BMD) Assessed by DXA
Description: The DXA BMD measures were assessed every 6 months over 5 years, and at a follow-up visit post-HPTH therapy. Due to varying lengths of time on each participant was on HPTH, these BMD assessment times were collapsed for purposes of analysis to: baseline, 6-month on HPTH therapy, last visit on HPTH therapy, and the post-HPTH follow-up visit. The Whole Body BMD is one of 6 bone regions measurements of bone mineralization density assessed by DXA.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
g/cm^2
  Raw BMD at Baseline | 1.248 (0.0162)
  Raw BMD at 6 months | 1.230 (0.0198)
  Raw BMD at last HPTH visit: number analyzed (Participants) | 17
  Raw BMD at last HPTH visit | 1.193 (0.0213)
  Raw BMD at Follow-up: number analyzed (Participants) | 17
  Raw BMD at Follow-up | 1.228 (0.0241)

41. Secondary Outcome: Perceived Interference (PI) of the Fatigue Symptom Inventory (FSI)
Description: Perceived interference is measured using seven separate items that assess the degree to which fatigue in the past week was judged to interfere with general level of activity, ability to bathe and dress, normal work activity, ability to concentrate, relations with others, enjoyment of life, and mood. The interference ratings were summed to yield a total interference score ranging from 0 (no perceived interference due to fatigue) to 70 (maximum possible perceived interference due to fatigue).
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
score on a scale
  Baseline visit | 18.9 (3.40)
  Six-month visit after start of HPTH | 15.3 (3.20)
  Last visit on HPTH prior to weaning: number analyzed (Participants) | 22
  Last visit on HPTH prior to weaning | 15.6 (3.74)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 19.3 (4.45)

42. Secondary Outcome: Average Severity Score of the Fatigue Symptom Inventory (FSI)
Description: Severity is measured using four separate items of the FSI questionnaire that assesses how the participant felt on their most, least, and average fatigue days in the past week as well as current fatigue. Participants score their level of fatigue for each item on an 11-point scale (0=not at all fatigued, 10=as fatigued as I could be). An average is taken of sum of these 4 scores. The average severity score can range from 0 to 10. A higher average severity score indicates that the participant is experiencing more severe fatigue.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
score on a scale
  Baseline visit | 4.16 (0.398)
  Six-month visit after start of HPTH | 3.53 (0.356)
  Last visit on HPTH prior to weaning: number analyzed (Participants) | 22
  Last visit on HPTH prior to weaning | 3.63 (0.427)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 4.03 (0.638)

43. Secondary Outcome: Composite Severity Score of the Fatigue Symptom Inventory (FSI)
Description: Severity is measured using four separate items of the FSI questionnaire that assesses how the participant felt on their most, least, and average fatigue days in the past week as well as current fatigue. Participants score their level of fatigue for each item on an 11-point scale (0=not at all fatigued, 10=as fatigued as I could be). The composite severity score reflects the sum of these 4 scores. The composite severity scores can range from 0 to 40. A higher composite severity scores indicates that the participant is experiencing more severe fatigue.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: Composite score from the FSI
Groups:
- Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined: Cohort 1 consisted of previously enrolled participants who were on HPTH therapy, were re-consented, and allowed to continue on the current study as a separate group. These participants were not randomized to a bone biopsy year, nor did they have additional biopsies performed. Cohort 1 participants were followed for safety outcomes only. Cohort 2 were previously enrolled participants on conventional care, were re-consented, re-enrolled, and randomized to a biopsy year. Cohort 3 consisted of all new participants consent, enrolled and randomized to a biopsy year. Efficacy outcomes were only analyzed for Cohorts 2 and 3 combined.
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
Composite score from the FSI
  Baseline visit | 15.4 (1.56)
  Six-month visit after start of HPTH | 14.1 (1.43)
  Last visit on HPTH prior to weaning: number analyzed (Participants) | 22
  Last visit on HPTH prior to weaning | 14.6 (1.69)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 16.1 (2.55)

44. Secondary Outcome: Total Distance Walked During a 6-minute Walk
Description: The total distance a participant was able to walk during a 6-minute walk
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: Distance in meters
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
Distance in meters
  Baseline visit | 606.3 (19.50)
  Six-month visit after start of HPTH: number analyzed (Participants) | 23
  Six-month visit after start of HPTH | 608.0 (18.83)
  Last visit on HPTH prior to weaning: number analyzed (Participants) | 22
  Last visit on HPTH prior to weaning | 567.2 (23.16)
  Post-HPTH follow-up visit: number analyzed (Participants) | 17
  Post-HPTH follow-up visit | 604.5 (26.67)

45. Secondary Outcome: SF36 Bodily Pain Domain
Description: The Bodily Pain (BP) domain scores are derived from the SF36 Health Survey taken by the participant. The SF-36 is a validated questionnaire assessing 4 physical domains: physical function, physical role limitations, bodily pain, and general health, and 4 mental domains: vitality, emotional role limitations, social function and mental health. From the 36 questions asked, a scoring tool derives SF36 domain scores for each of the eight domains. These domain scores are scaled to range from 0 to 100 with a population mean of 50 and a standard deviation of 10. Lower scores indicate more disability; and, higher scores indicate less disability. The BP domain scores indicate to what extent a participant's bodily pain hinders their performance of daily activities.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
score on a scale
  Baseline visit | 48.97 (1.749)
  Six-month visit after start of HPTH | 49.53 (1.705)
  Last visit on HPTH prior to weaning | 47.52 (1.628)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 47.02 (2.709)

46. Secondary Outcome: SF36 Emotional Role Limitations Domain
Description: Emotional Role Limitations (RE) Domain scores are derived from the SF36 Health Survey taken by the participant. The SF-36 is a validated questionnaire assessing 4 physical domains: physical function, physical role limitations, bodily pain, and general health, and 4 mental domains: vitality, emotional role limitations, social function and mental health. From the 36 questions asked, a scoring tool derives SF36 domain scores for each of the eight domains. These domain scores are scaled to range from 0 to 100 with a population mean of 50 and a standard deviation of 10. Lower scores indicate more disability; and, higher scores indicate less disability. The RE Domain score assesses the extent to which the emotional condition of the participant, e.g. feeling depressed or anxious, limits his/her daily functioning and ability to perform roles, such as in cutting down on the amount of time spent on work or other activities and accomplishing less than he/she would like to.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
score on a scale
  Baseline visit | 48.27 (2.310)
  Six-month visit after start of HPTH | 51.34 (1.852)
  Last visit on HPTH prior to weaning | 51.02 (1.539)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 47.24 (3.040)

47. Secondary Outcome: SF36 General Health Domain
Description: General Health (GH) Domain scores are derived from the SF36 Health Survey taken by the participant. The SF-36 is a validated questionnaire assessing 4 physical domains: physical function, physical role limitations, bodily pain, and general health, and 4 mental domains: vitality, emotional role limitations, social function and mental health. From the 36 questions asked, a scoring tool derives SF36 domain scores for each of the eight domains. These domain scores are scaled to range from 0 to 100 with a population mean of 50 and a standard deviation of 10. Lower scores indicate more disability; and, higher scores indicate less disability. The GH domain score assesses a participant's perception of their general health in terms of concepts such as excellent, very good, good, fair or poor, getting ill easier than other people, and just as healthy as anyone he/she knows.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
score on a scale
  Baseline visit | 43.80 (1.907)
  Six-month visit after start of HPTH | 48.11 (1.801)
  Last visit on HPTH prior to weaning | 45.25 (1.976)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 42.45 (2.578)

48. Secondary Outcome: SF36 Mental Health Domain
Description: Mental Health (MH) Domain scores are derived from the SF36 Health Survey taken by the participant. The SF-36 is a validated questionnaire assessing 4 physical domains: physical function, physical role limitations, bodily pain, and general health, and 4 mental domains: vitality, emotional role limitations, social function and mental health. From the 36 questions asked, a scoring tool derives SF36 domain scores for each of the eight domains. These domain scores are scaled to range from 0 to 100 with a population mean of 50 and a standard deviation of 10. Lower scores indicate more disability; and, higher scores indicate less disability. The MH domain assesses the extent to which the participant is, among other things, feeling full of pep, is happy, is feeling calm and peaceful, is very nervous, or is feeling worn out and tired.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
score on a scale
  Baseline visit | 47.07 (2.120)
  Six-month visit after start of HPTH | 49.51 (1.736)
  Last visit on HPTH prior to weaning | 49.30 (2.029)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 47.04 (2.793)

49. Secondary Outcome: SF36 Physical Function Domain
Description: Physical Function (PF) Domain scores are derived from the SF36 Health Survey taken by the participant. The SF-36 is a validated questionnaire assessing 4 physical domains: physical function, physical role limitations, bodily pain, and general health, and 4 mental domains: vitality, emotional role limitations, social function and mental health. From the 36 questions asked, a scoring tool derives SF36 domain scores for each of the eight domains. These domain scores are scaled to range from 0 to 100 with a population mean of 50 and a standard deviation of 10. Lower scores indicate more disability; and, higher scores indicate less disability. The PF domain assesses the extent to which the participant's perceptions of his/her ability to perform vigorous and moderate physical activities are influenced by his/her physical condition.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
score on a scale
  Baseline visit | 49.14 (1.479)
  Six-month visit after start of HPTH | 51.07 (1.265)
  Last visit on HPTH prior to weaning | 48.97 (1.807)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 47.91 (2.333)

50. Secondary Outcome: SF36 Physical Role Limitations Domain
Description: Physical Role Limitations (RP) Domain scores are derived from the SF36 Health Survey taken by the participant. The SF-36 is a validated questionnaire assessing 4 physical domains: physical function, physical role limitations, bodily pain, and general health, and 4 mental domains: vitality, emotional role limitations, social function and mental health. From the 36 questions asked, a scoring tool derives SF36 domain scores for each of the eight domains. These domain scores are scaled to range from 0 to 100 with a population mean of 50 and a standard deviation of 10. Lower scores indicate more disability; and, higher scores indicate less disability. The RP Domain assesses the extent to which a participant's' performance of his/her roles in daily activities is impeded by his/her physical state of health.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
score on a scale
  Baseline visit | 44.10 (2.085)
  Six-month visit after start of HPTH | 45.73 (2.206)
  Last visit on HPTH prior to weaning | 48.49 (1.699)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 45.56 (2.938)

51. Secondary Outcome: SF36 Social Function Domain
Description: Social Function (SF) Domain scores are derived from the SF36 Health Survey taken by the participant. The SF-36 is a validated questionnaire assessing 4 physical components: physical function, physical role limitations, bodily pain, and general health, and 4 mental components: vitality, emotional role limitations, social function and mental health. From the 36 questions asked, a scoring tool is used to calculate each of the eight domain scores. The scoring tool transforms the score into a 0-100 scale on the assumption that each question carries equal weight. SF36 domain scores are scaled to have a population mean of 50 and a standard deviation of 10. The SF Domain assesses the level of a participant's social activities and interaction with significant others such as family members, friends, neighbours and other social relations. Lower scores indicate more disability; higher scores indicate less disability with respect to social function.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
score on a scale
  Baseline visit | 46.40 (2.562)
  Six-month visit after start of HPTH | 48.67 (2.178)
  Last visit on HPTH prior to weaning | 49.12 (2.048)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 42.00 (2.782)

52. Secondary Outcome: SF36 Vitality Domain
Description: Vitality (VT) Domain scores are derived from the SF36 Health Survey taken by the participant. SF36 domain scores are scaled to have a population mean of 50 and a standard deviation of 10. Higher scores reflect a better quality of life.The SF-36 is a validated questionnaire assessing 4 physical components: physical function, physical role limitations, bodily pain, and general health, and 4 mental components: vitality, emotional role limitations, social function and mental health. From the 36 questions asked, a scoring tool is used to calculate the eight domain scores. The scoring tool transforms the score into a 0-100 scale on the assumption that each question carries equal weight. SF36 domain scores are scaled to have a population mean of 50 and a standard deviation of 10. Lower scores indicate more disability; and, higher scores indicate less disability. The VT Domain assesses the participant's experience of feeling energetic and full of pep, or worn out and tired.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
score on a scale
  Baseline visit | 43.37 (2.347)
  Six-month visit after start of HPTH | 46.89 (2.090)
  Last visit on HPTH prior to weaning | 48.45 (2.284)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 44.98 (2.457)

53. Secondary Outcome: Serum Alkaline Phosphatase
Description: Serum Alkaline Phosphatase concentration
Time Frame: Baseline, last visit on HPTH (up to 5 years), and post-HPTH follow-up visit (6 months post last visit on HPTH)
Population: as for outcome 35
Measure: Mean (Standard Error); unit: ug/L
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
ug/L
  Baseline visit | 9.92 (1.017)
  Last visit on HPTH prior to weaning: number analyzed (Participants) | 22
  Last visit on HPTH prior to weaning | 33.34 (5.148)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 12.69 (3.254)

54. Secondary Outcome: Serum Calcium
Description: Serum Calcium concentration
Time Frame: Baseline, last visit on HPTH (up to 5 years), and post-HPTH follow-up visit (6 months post last visit on HPTH)
Population: as for outcome 35
Measure: Mean (Standard Error); unit: Mmol/L
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
Mmol/L
  Baseline visit | 2.02 (0.035)
  Last visit on HPTH prior to weaning: number analyzed (Participants) | 22
  Last visit on HPTH prior to weaning | 2.06 (0.028)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 2.02 (0.041)

55. Secondary Outcome: Serum Osteocalcin
Description: Serum Osteocalcin concentration
Time Frame: Baseline, last visit on HPTH (up to 5 years), and post-HPTH follow-up visit (6 months post last visit on HPTH)
Population: as for outcome 35
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
ng/mL
  Baseline visit | 14.86 (0.877)
  Last visit on HPTH prior to weaning: number analyzed (Participants) | 22
  Last visit on HPTH prior to weaning | 164.6 (28.390)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 49.15 (22.412)

56. Secondary Outcome: Serum Phosphorus
Description: Serum Phosphorus concentration
Time Frame: Baseline, last visit on HPTH (up to 5 years), and post-HPTH follow-up visit (6 months post last visit on HPTH)
Population: as for outcome 35
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
mg/dL
  Baseline visit | 4.74 (0.118)
  Last visit on HPTH prior to weaning: number analyzed (Participants) | 22
  Last visit on HPTH prior to weaning | 4.62 (0.108)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 4.59 (0.145)

57. Secondary Outcome: 24 Hour Urine NTX Telopeptide
Description: Urine was collected over 24 hours and the total NTX Telopeptide measured
Time Frame: Baseline, last visit on HPTH (up to 5 years), and post-HPTH follow-up visit (6 months post last visit on HPTH)
Population: as for outcome 35
Measure: Mean (Standard Error); unit: nmol Bone Collagen Equiv/mmol Creatinine
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
nmol Bone Collagen Equiv/mmol Creatinine
  Baseline visit | 21.35 (6.117)
  Last visit on HPTH prior to weaning: number analyzed (Participants) | 22
  Last visit on HPTH prior to weaning | 305.1 (60.885)
  Post-HPTH follow-up visit: number analyzed (Participants) | 18
  Post-HPTH follow-up visit | 29.89 (14.758)

58. Secondary Outcome: Number of Participants With Nephrolithiasis/Nephrocalcinosis
Description: Participants had ultrasound and CT imaging of the kidney were performed yearly. The rates of new, stable, and progressing nephrocalcinosis and nephrolithiasis (NCNL) were recorded.
Time Frame: Baseline, 12-Month Visit, 24-Month Visit, 36-Month Visit, 48-Month Visit, and 60-Month Visit
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
Participants
  No detectable NCNL at any time during study | 5
  Baseline NCNL that remains stable on HPTH therapy | 7
  New/progressing NCNL on HPTH therapy | 10
  NCNL that resolved on HPTH therapy | 2

59. Secondary Outcome: Primary Bone Biopsy Measures Adjusted for HPTH Dose
Description: The 8 primary bone biopsy measures were to be adjusted HPTH dose by fitting the primary bone biopsy model with both linear and quadratic dose covariates added to the model. However, the study was terminated early resulting in only 5, 5, and 2 participants having their biopsies at 1, 2, and 4 years respectively. To add additional linear and quadratic dose covariates to the statistical model with an already small sample sizes would highly risk over-parameterizing the model. Thus no new analysis was performed.
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 0

60. Secondary Outcome: Sensitivity Analyses of Female Menopause Status in the Primary Bone Biopsy Efficacy Models
Description: As a sensitivity analysis, the 8 primary bone biopsy measures were to be adjusted for female menopausal status, by fitting the primary bone biopsy model with a menopausal status covariate added to the model. However, the study was terminated early resulting in only 5, 5, and 2 participants having their biopsies at 1, 2, and 4 years respectively. Furthermore, 3 males would need to be removed from the model leaving 4, 3, 2 participants with bone biopsies with an additional degree of freedom consumed for the menopausal status covariate. Thus, the planned mixed models analysis was not performed since with such small samples sizes random fluctuations in the data could give misleading erroneous results.
Time Frame: Baseline, 1 year bone biopsy, and combined 2 and 4 year bone biopsies
Population: as for outcome 1
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 0

61. Secondary Outcome: Z-score of 1/3 Radius Bone Mineralization Density (BMD) Assessed by DXA.
Description: The DXA BMD measures were assessed every 6 months over 5 years, and at a follow-up visit post-HPTH therapy. Due to varying lengths of time on each participant was on HPTH, these BMD assessment times were collapsed for purposes of analysis to: baseline, 6-month on HPTH therapy, last visit on HPTH therapy, and the post-HPTH follow-up visit The 1/3 Radius BMD is one of 6 bone regions measurements of bone mineralization density assessed by DXA. The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
z-score
  Z-score BMD at Baseline | 0.89 (0.197)
  Z-score BMD at 6 months | 0.82 (0.190)
  Z-score BMD at last HPTH visit: number analyzed (Participants) | 17
  Z-score BMD at last HPTH visit | 0.26 (0.273)
  Z-score BMD at Follow-up: number analyzed (Participants) | 18
  Z-score BMD at Follow-up | 0.50 (0.276)

62. Secondary Outcome: Z-score of AP Spine Bone Mineralization Density (BMD) Assessed by DXA
Description: The DXA BMD were assessed every 6 months over 5 years, and at a follow-up visit post-HPTH therapy. Due to varying lengths of time on each participant was on HPTH, these BMD assessment times were collapsed for purposes of analysis to: baseline, 6-month on HPTH therapy, last visit on HPTH therapy, and the post-HPTH follow-up visit. The AP Spine BMD is one of 6 bone regions measurements of bone mineralization density assessed by DXA. The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes.
Time Frame: Baseline, 6-months after start of HPTH, last visit on HPTH, and post-HPTH follow-up visits
Population: as for outcome 35
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
z-score
  Z-score BMD at Baseline | 1.46 (0.221)
  Z-score BMD at 6 months | 1.15 (0.207)
  Z-score BMD at last HPTH visit: number analyzed (Participants) | 17
  Z-score BMD at last HPTH visit | 1.24 (0.279)
  Z-score BMD at Follow-up: number analyzed (Participants) | 18
  Z-score BMD at Follow-up | 2.30 (0.306)

63. Secondary Outcome: Z-score of Femoral Neck Bone Mineralization Density (BMD) Assessed by DXA
Description: The DXA BMD measures were assessed every 6 months over 5 years, and at a follow-up visit post-HPTH therapy. Due to varying lengths of time on each participant was on HPTH, these BMD assessment times were collapsed for purposes of analysis to: baseline, 6-month on HPTH therapy, last visit on HPTH therapy, and the post-HPTH follow-up visit. The Femoral BMD is one of 6 bone regions measurements of bone mineralization density assessed by DXA. The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes.
Time Frame: Baseline, 6-months after start of HPTH, last visit on HPTH, and post-HPTH follow-up visits
Population: as for outcome 35
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
z-score
  Z-score BMD at Baseline | 0.85 (0.192)
  Z-score BMD at 6 months | 0.59 (0.186)
  Z-score BMD at last HPTH visit: number analyzed (Participants) | 17
  Z-score BMD at last HPTH visit | 0.99 (0.229)
  Z-score BMD at Follow-up: number analyzed (Participants) | 18
  Z-score BMD at Follow-up | 1.10 (0.249)

64. Secondary Outcome: Z-score of Lateral Spine Bone Mineralization Density (BMD) Assessed by DXA
Description: The DXA BMD were assessed every 6 months over 5 years, and at a follow-up visit post-HPTH therapy. Due to varying lengths of time on each participant was on HPTH, these BMD assessment times were collapsed for purposes of analysis to: baseline, 6-month on HPTH therapy, last visit on HPTH therapy, and the post-HPTH follow-up visit. The Lateral Spine BMD is one of 6 bone regions measurements of bone mineralization density assessed by DXA . The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes.
Time Frame: Baseline, 6-months after start of HPTH, last visit on HPTH, and post-HPTH follow-up visits
Population: as for outcome 35
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
z-score
  Z-score BMD at Baseline: number analyzed (Participants) | 15
  Z-score BMD at Baseline | 2.16 (0.215)
  Z-score BMD at 6 months: number analyzed (Participants) | 16
  Z-score BMD at 6 months | 2.22 (0.223)
  Z-score BMD at last HPTH visit: number analyzed (Participants) | 12
  Z-score BMD at last HPTH visit | 3.87 (0.483)
  Z-score BMD at Follow-up: number analyzed (Participants) | 13
  Z-score BMD at Follow-up | 4.72 (0.737)

65. Secondary Outcome: Z-score of Total Hip Bone Mineralization Density (BMD) Assessed by DXA
Description: The DXA BMD measures were assessed every 6 months over 5 years, and at a follow-up visit post-HPTH therapy. Due to varying lengths of time on each participant was on HPTH, these BMD assessment times were collapsed for purposes of analysis to: baseline, 6-month on HPTH therapy, last visit on HPTH therapy, and the post-HPTH follow-up visit. The Total Hip BMD is one of 6 bone regions measurements of bone mineralization density assessed by DXA. The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes.
Time Frame: Baseline, 6-months after start of HPTH, last visit on HPTH, and post-HPTH follow-up visits
Population: as for outcome 35
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
z-score
  Z-score BMD at Baseline | 0.85 (0.161)
  Z-score BMD at 6 months | 0.66 (0.165)
  Z-score BMD at last HPTH visit: number analyzed (Participants) | 17
  Z-score BMD at last HPTH visit | 0.89 (0.212)
  Z-score BMD at Follow-up: number analyzed (Participants) | 18
  Z-score BMD at Follow-up | 1.01 (0.172)

66. Secondary Outcome: Z-score of Whole Body Bone Mineralization Density (BMD) Assessed by DXA
Description: The DXA BMD measures were assessed every 6 months over 5 years, and at a follow-up visit post-HPTH therapy. Due to varying lengths of time on each participant was on HPTH, these BMD assessment times were collapsed for purposes of analysis to: baseline, 6-month on HPTH therapy, last visit on HPTH therapy, and the post-HPTH follow-up visit. The Whole Body BMD is one of 6 bone regions measurements of bone mineralization density assessed by DXA. The unit of measure is a z-score. Z-scores are normed to standard populations to a mean of zero and a standard deviation of 1. The normal range for a z-score is from -2 to 2. Values above or below this normal range are considered worse outcomes.
Time Frame: Baseline, 6-months after start of HPTH, last visit on HPTH, and post-HPTH follow-up visits
Population: as for outcome 35
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Cohorts 2 (CC on Old Study) and 3 (Newly Enrolled) Combined
Number analyzed (Participants) | 24
z-score
  Z-score BMD at Baseline: number analyzed (Participants) | 20
  Z-score BMD at Baseline | 1.59 (0.193)
  Z-score BMD at 6 months: number analyzed (Participants) | 20
  Z-score BMD at 6 months | 1.32 (0.180)
  Z-score BMD at last HPTH visit: number analyzed (Participants) | 17
  Z-score BMD at last HPTH visit | 0.66 (0.172)
  Z-score BMD at Follow-up: number analyzed (Participants) | 17
  Z-score BMD at Follow-up | 1.12 (0.173)

ADVERSE EVENTS:
Time Frame: From time of the start of HPTH therapy through the date of last dose of HPTH (i.e., the end of the weaning period off HPTH). The last dose occurred up to 64 months after the start of HPTH therapy.
Description: Treatment emergent adverse events are those events that begin on or after the first dose of HPTH through the date last dose of HPTH.
Groups:
- All Cohorts, Treated With HPTH on the New Study: Participants from Cohorts 1, 2, and 3, who were treated with HPTH on the new study.
Arm/Group | All Cohorts, Treated With HPTH on the New Study
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 8/31
Other Adverse Events (participants affected / at risk) | 28/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Cohorts, Treated With HPTH on the New Study (N=31)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (7)
Headache (Nervous system disorders) | 1 (1)
Hypocalcaemic seizure (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Cohorts, Treated With HPTH on the New Study (N=31)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Coeliac disease (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival disorder (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (7)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (10)
Chest pain (General disorders) | 1 (1)
Chronic fatigue syndrome (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Injection site dryness (General disorders) | 1 (1)
Injection site erythema (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 3 (4)
Ear infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Herpes zoster (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 7 (8)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4)
Urinary tract infection (Infections and infestations) | 4 (6)
Viral infection (Infections and infestations) | 3 (3)
Wound infection (Infections and infestations) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 4 (4)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision site pruritus (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 2 (3)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Bone density decreased (Investigations) | 2 (2)
Cardiac murmur (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 2 (2)
Weight decreased (Investigations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (10)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 4 (4)
Hyperreflexia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2)
Thoracic outlet syndrome (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Flank pain (Renal and urinary disorders) | 2 (2)
Hypocitraturia (Renal and urinary disorders) | 15 (16)
Micturition urgency (Renal and urinary disorders) | 3 (3)
Nephrocalcinosis (Renal and urinary disorders) | 6 (6)
Nephrolithiasis (Renal and urinary disorders) | 14 (14)
Pollakiuria (Renal and urinary disorders) | 3 (3)
Renal cyst (Renal and urinary disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (4)
Varicose vein (Vascular disorders) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT00395538/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2015-09-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT00395538/Prot_ICF_001.pdf